CLINICAL TRIAL: NCT00205855
Title: Stimulus Confirmatory Study - An Implantable Spinal Cord Stimulation Pain Management System
Brief Title: An Implantable Spinal Cord Stimulation Pain Management System
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-S-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Pain; Pain, Intractable; Pain; Back Pain; Failed Back Surgery Syndrome
Keywords: Pain; Chronic Pain; Neurostimulation
MeSH Terms: conditions — Chronic Pain; Pain, Intractable; Pain; Back Pain; Failed Back Surgery Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Precision SCS (Experimental): Precision SCS. Patients who receive Precision Spinal Cord Stimulator (SCS) Stimulus system
  Interventions: Device: Precision SCS

INTERVENTIONS:
Device: Precision SCS — Advanced Bionics totally implantable Spinal Cord Stimulation (SCS) System, the Stimulus System. This system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: failed back surgery syndrome, intractable low back pain and leg pain.
  Other Names: Stimulus System; PRECISION Spinal Cord Stimulator System (PRECISION System)

SUMMARY:
There are many treatment options available for the management of chronic pain . Some include, but are not limited to, over-the-counter medications, Non-Steroidal Anti-Inflammatory Drugs, Physical Therapy, Transcutaneous Electrical Nerve Stimulation (TENS) and nerve blocks. Historically, the mainstay of pain treatment has been pharmacotherapy. However, pharmacotherapy has varying degrees of effectiveness and is often associated with undesirable side effects. Although many patients are successfully treated, for those who fail some of these more conservative therapies the remaining option is limited to spinal cord stimulation (SCS), proven to be an effective therapy to more than half of those failing conservative treatments . Over 50% of those who have failed these more conservative methods of pain management, can now, under the guidance of a clinician utilizing SCS, have their pain levels successfully managed. SCS is a less invasive therapy that is a reversible treatment with greater long-term benefits than more permanent, radical approaches and one that deserves greater consideration in the management of chronic, intractable pain.

DETAILED DESCRIPTION:
This clinical trial was a confirmatory study for the Advanced Bionics totally implantable Spnial Cord Stimulation(SCS) System, the Stimulus System. This system is indicated as an aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with the following: Dailed back surgery syndrome, intractable low backpain and leg pain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with chronic, intractable pain of the trunk and/or limbs which includes but is not limited to, unilateral or bilateral pain associated with any of the following: failed back surgery syndrome, intractable low back pain and leg pain.
2. Be an appropriate candidate for surgery.
3. Be capable of giving informed consent.
4. Be capable and willing to follow all study related procedures.

Exclusion Criteria:

1. Have an inability to operate the system either by self or care-giver.
2. Are currently participating or have participated within the past 30 days in any clinical investigation that could conflict with the requirements of this study.
3. Have any implanted electrical devices, regardless of whether active or inactive.
4. Have any active implantable device regardless of whether stimulation is ON or OFF.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-02; Primary Completion 2003-10 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kay Adair, Study Chair — Boston Scientific Corporation
Locations (9):
- United States (9):
  - Alabama Pain Center, Huntsville, Alabama
  - California Pain Medicine Centers, Los Angeles, California
  - Pacific Pain Treatment Center, San Francisco, California
  - Yellowstone Neurological Associates, Billings, Montana
  - Northshore University Hospital, Syosset, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Dallas Neurological Associates, Dallas, Texas
  - River Oaks Pain Management, Houston, Texas
  - Texas Back Institute, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Spinal Cord Stimulation (SCS) Group: Upon meeting entry criteria and a baselineline evaluation all eligible subjects then receive either a temporary lead or a permanent lead (both leads are considered "trial" durign this phase) attached to an external stimulator for a minimum period of 48 hours. Patients who are determined to have 50% improvement in the VAS score from baseline after the trial phase were implanted with the Precision Spinal Cord Stimulation System.
Period: Overall Study
Arm/Group | Spinal Cord Stimulation (SCS) Group
Started | 65
Completed | 44
Not Completed | 21
Not completed — Only received temporary implants | 16
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Groups:
- Spinal Cord Stimulation (SCS) Group: Precision Spinal Cord Stimulation therapy group
Arm/Group | Spinal Cord Stimulation (SCS) Group
Number analyzed (Participants) | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Score From Baseline to 2 Week Post Initial Fitting.
Description: The VAS score is rated by the patient for the average pain level within the past 7 days where on a scale of 0 to 10, 0 is equal to"no pain" and 10 is equal to "worst pain imaginable." This measurement is captured at baseline and again at 2 weeks post intitial fitting. The measurement is the percent difference between the VAS at 2 weeks post intital fitting from the baseline VAS.
Time Frame: 2 weeks post initial fitting
Measure: Number; unit: participants with > 50% VAS improvement
Arm/Group | Spinal Cord Stimulation (SCS) Group
Number analyzed (Participants) | 46
participants with > 50% VAS improvement | 35

ADVERSE EVENTS:
Arm/Group | Spinal Cord Stimulation (SCS) Group
Serious Adverse Events (participants affected / at risk) | 12/65
Other Adverse Events (participants affected / at risk) | 20/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (SCS) Group (N=65)
Lead Migration (Surgical and medical procedures) | 5 (5)
Loss of Therapy (Surgical and medical procedures) | 1 (1)
New Lead Placement (Surgical and medical procedures) | 2 (2)
Infection (Infections and infestations) | 2 (2)
Implantable Pulse Generator Movement (Surgical and medical procedures) | 1 (1)
Pain (Surgical and medical procedures) | 1 (1)
Device Malfunction (Surgical and medical procedures) | 1 (1)
Death (Musculoskeletal and connective tissue disorders) | 1 (1) — Died in t he hospital due to complications of a broken hip
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Spinal Cord Stimulation (SCS) Group (N=65)
Abstinence syndrome (Nervous system disorders) | 1 (1)
CSF leak (Injury, poisoning and procedural complications) | 3 (3)
Infection (Infections and infestations) | 1 (1)
Lead Migration (Surgical and medical procedures) | 4 (4)
Device Malfunction (Injury, poisoning and procedural complications) | 8 (8)
Grand-Mal Seizure (Nervous system disorders) | 1 (1)
Nausea & Vomiting (Gastrointestinal disorders) | 1 (1)
Reduced Telemetry Range (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Pain during SCS Trial (Injury, poisoning and procedural complications) | 1 (1)
Over and Under stimulation during SCS Trial (Injury, poisoning and procedural complications) | 4 (4)
Unpleasant Stimulation (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less